CLINICAL TRIAL: NCT05788523
Title: Prediction Of Serious Adverse Event in Emergency Department With dysKAlemia, Retrospective Study
Acronym: PODKA-R
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Collaborators: Georgia Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-01Obs-CHRMT
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-02

CONDITIONS: Emergencies
Keywords: artificial intelligence; kalemia; dyskalemia
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dyskalemia, hypo- and hyperkalemia are common in the emergency department and are associated with increased morbidity and mortality.

The potential seriousness of dyskalemia results from the potential alteration of intracardiac conduction and the increase in cardiac rhythm disorders, all associated with a lethal risk. Given the aspecific symptoms of dyskalemia and the complex causal links to be acquired, it is difficult to judge the severity of the disorders in front of an initial clinical presentation of a patient in the emergency room, as the patient may present a serious condition during his stay in the emergency room, related to the dyskalemia and not prejudged at first. The ECG is recommended to judge the severity of the disorder, in association with the level of kalemia, but the electrical changes of its pattern in the context of dyskalemia are sometimes so fine that even the eye of the practitioner is not able to detect them. To date and to our knowledge, there is no tool for predicting the risk of RTA or death in dyskalemia. The existing studies on the subject, including ECGs, seek to detect dyskalemia and not its complications, and the proposed tools only take into account the ECG and not the clinical context of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Major patient consulting in an emergency department participating in the study
* who received at least a digital ECG AND an ionogram in the emergency department during the study period

Exclusion Criteria:

* Patient who has expressed opposition to the reuse of their data for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients consulted in the emergency unit of the participating centre, with quality criteria for the EHCs; this cohort will validate the Artificial Intelligence method developed in partnership with the laboratory
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with Cardiac arrest and/or rhythm disorder | within 48 hours
  Number of patients with Cardiac arrest and/or rhythm disorder within 48 hours of the ED visit

SECONDARY OUTCOMES:
Rate of Mortality | within 48 hours
  Rate of Mortality : all causes combined (SAU, hospitalization, SMUR, home)
The type of received treatment for dyskalemia | within 48 hours
  The type of treatment received for dyskalemia (IV and what type, orally and what type)

CONTACTS AND LOCATIONS:
Overall Officials: Laure ABENSUR VUILLAUME, MD, PhD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, France

IPD SHARING:
Plan to Share IPD: No